CLINICAL TRIAL: NCT04321187
Title: Influence of Radiotherapy on the Dynamics of Aging in Prostate Cancer Patients
Brief Title: Influence of Prostate Cancer Radiation on Aging
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 31-437 ex 18/19
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer; Aging Disorder; Radiotherapy; Complications; Inflammation
Keywords: telomere length; aging; radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ethylenediaminetetraacetic acid blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have reported that cancer survivors develop age-related chronic conditions like frailty, sarcopenia, cardiac dysfunction, and cognitive impairment earlier and/or at a greater burden than similarly aged individuals never diagnosed with cancer or exposed to cancer therapies.

However, the knowledge about aging-associated consequences of cancer treatment and the processes that underlie differential responses to therapy is very limited. In 2018, a think tank established by the National Cancer Institute has defined various research needs to expand the evidence base for aging-related consequences of cancer treatment, such as studies to examine aging-related processes that include regularly performed assessments capturing factors associated with physical function or studies to elucidate pathways that lead to the emergence of aging phenotypes and to understand the relationships between biomarkers of aging and functional outcomes in cancer survivors. In addition, study inclusion of older adults with comorbidities and higher levels of frailty has been proposed to achieve an improved understanding of functional outcomes at any age.

Hypotheses / objectives We hypothesize that prostate cancer radiotherapy accelerates aging-related processes, furthermore, aging-related biomarkers may predict functional outcomes and represent early indicators of aging phenotypes. Primary objectives of the proposed study are the determination of the aging-related consequences of radiotherapy in prostate cancer patients and the evaluation of the relationship between biomarkers of aging and age-related clinical conditions.

DETAILED DESCRIPTION:
Systematic evaluations of functional and cognitive status, comorbidities, health status, mobility, nutritional status, psychological status, and social circumstances as well as measurements of cellular senescence and chronic inflammation will be performed in a cohort of prostate cancer patients at baseline (before radiotherapy), at the end of radiotherapy and at follow-up intervals thereafter. The evaluation of aging-related biomarkers will include determination of markers of cellular senescence and markers of systemic inflammation. The correlation between genetic variants modulating telomere length and the risk of developing age-related phenotypes will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer
* Candidate to definitive radiation treatment
* Local or locally advanced disease
* Aged ≥ 65 years
* Informed consent

Exclusion Criteria:

* Unable to give written informed consent
* Metastatic disease

Ages: 70 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: prostate cancer patients treated at the Department of Therapeutic Radiology and Oncology, Comprehensive Cancer Center, Medical University of Graz. Prostate cancer patients who are candidates for curative radiotherapy will be invited to take part by the local investigators.
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Functionality - activities of daily living | 2 years
  Functional decline measured by Activities of Daily Living examination (range, 0-6; high values indicate high functionality and improved outcome)
Functionality - instrumental activities of daily living | 2 years
  Functional decline measured by the Instrumental Activities of Daily Living examination (range, 0-8; high values indicate high functionality and improved outcome)
Cognitive disorder | 2 years
  Cognitive disorder measured by the Mini-Mental State Examination (range, 0-30; high values indicate normal cognition and improved outcome)
Comorbidities | 2 years
  Comorbidities measured by the Charlson comorbidity index (range, 0-37; high score indicates high rate of comorbidities and worse outcome)
Mental disorder | 2 years
  Mental disorder measured by the Geriatric depression scale (range, 0-30; higher values indicate depression and worse outcome)
Mobility | 2 years
  Mobility measured by the Timed up and go test (≥12 seconds to complete the Timed up and go test indicates mobility impairment and worse outcome)
Number of medications taken | 2 years
  Polypharmacy represents an aging related condition (high number of medication taken indicates worse outcome)

SECONDARY OUTCOMES:
Radiation induced toxicity | 10 years
  Frequency of acute and late side effects

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Langsenlehner, Principal Investigator — Medical University of Graz, Dept. of Therapeutic Radiology and Oncology
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
In is not planned to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Renner W, Krenn-Pilko S, Gruber HJ, Herrmann M, Langsenlehner T. Relative telomere length and prostate cancer mortality. Prostate Cancer Prostatic Dis. 2018 Nov;21(4):579-583. doi: 10.1038/s41391-018-0068-3. Epub 2018 Aug 6. PMID 30082901
- [Background] Guida JL, Ahles TA, Belsky D, Campisi J, Cohen HJ, DeGregori J, Fuldner R, Ferrucci L, Gallicchio L, Gavrilov L, Gavrilova N, Green PA, Jhappan C, Kohanski R, Krull K, Mandelblatt J, Ness KK, O'Mara A, Price N, Schrack J, Studenski S, Theou O, Tracy RP, Hurria A. Measuring Aging and Identifying Aging Phenotypes in Cancer Survivors. J Natl Cancer Inst. 2019 Dec 1;111(12):1245-1254. doi: 10.1093/jnci/djz136. PMID 31321426